CLINICAL TRIAL: NCT06702787
Title: Mechanical Thrombectomy in the Middle East and North Africa: Interim Results from the MEMENTO Registry
Acronym: MEMENTO Regist
Status: Enrolling by invitation | Type: Observational
Sponsor: Middle East North Africa Stroke and Interventional Neurotherapies Organization (Other)
Responsible Party: Sponsor
Other Study IDs: MENASINO1002
Record Dates: First submitted 2024-11-14; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Stroke Acute; Endovascular Procedures; Large Vessel Occlusion
Keywords: Mechanical Thrombectomy; Acute Ischemic; Stroke Large Vessel Occlusion; Middle East and North Africa MENA Region; Endovascular Treatment; Cerebral Infarction; Brain Ischemia; Stroke Management; Reperfusion Therapy; Neurointervention Cerebrovascular
MeSH Terms: conditions — Stroke; Cerebral Infarction; Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The MEMENTO (MEchanical thrMobectomy NETwork for MENA TOgether) Registry is a multicenter, prospective observational study aiming to evaluate the effectiveness, safety, and cost-effectiveness of mechanical thrombectomy (MT) in patients with acute ischemic stroke (AIS) due to large vessel occlusions (LVO) in the Middle East and North Africa (MENA) region. This interim analysis reports on the first 499 patients enrolled, assessing clinical outcomes, procedural details, and economic implications.

DETAILED DESCRIPTION:
Detailed Description Stroke is a leading cause of morbidity and mortality worldwide, with a significant burden in the MENA region due to limited access to advanced stroke care therapies like mechanical thrombectomy (MT). The MEMENTO Registry seeks to collect real-world data on MT practices, outcomes, and accessibility in the MENA region to inform clinical practice and policy. The study includes AIS patients who underwent MT for confirmed LVO or medium vessel occlusion (MeVO), with or without prior intravenous thrombolysis (IV tPA), regardless of age, baseline NIHSS score, or time from symptom onset.

Data collected encompass demographics, clinical characteristics, imaging findings, procedural details, outcomes at discharge and follow-up, complications, and a cost-effectiveness analysis comparing MT to standard medical care (SMC). The primary outcome is functional independence at 90 days post-procedure, defined as a modified Rankin Scale (mRS) score of 0-2.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years and older (no upper age limit). Diagnosed with acute ischemic stroke due to confirmed large vessel occlusion (LVO) or medium vessel occlusion (MeVO).

Underwent mechanical thrombectomy (MT) with or without prior intravenous thrombolysis (IV tPA).

Pre-stroke modified Rankin Scale (mRS) score of 0-5. Consent to participate in the registry (by patient or legal representative).

Exclusion Criteria:

Absence of confirmed LVO or MeVO. Pre-stroke mRS score of 6. Known severe comorbid conditions precluding MT. Inability to obtain informed consent. Patients not treated with MT.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients presenting with acute ischemic stroke due to LVO or MeVO at participating centers in the MENA region, who received MT as part of standard clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-04-11 (Estimated); Study Completion 2025-09-11 (Estimated)

PRIMARY OUTCOMES:
Functional Independence at 90 Days | 90 days post-procedure
  Description: Proportion of patients achieving a modified Rankin Scale (mRS) score of 0-2 at 90 days post-procedure.

SECONDARY OUTCOMES:
Proportion of Patients Achieving TICI Score ≥2b After MT | Immediately post-procedure
  Proportion of patients achieving Thrombolysis in Cerebral Infarction (TICI) score ≥2b after MT.
  Scale Title: Thrombolysis in Cerebral Infarction (TICI) score Scale Range: 0 to 3 Outcome Interpretation: Higher scores indicate better outcomes, with a score of ≥2b representing successful reperfusion.
Improvement in NIHSS Score from Baseline to 24 Hours and at Follow-up | Baseline, 24 hours, and up to 90 days
  Improvement in National Institutes of Health Stroke Scale (NIHSS) score from baseline to 24 hours and at follow-up.
  Scale Title: National Institutes of Health Stroke Scale (NIHSS) Scale Range: 0 to 42 Outcome Interpretation: Lower scores indicate better outcomes, with a decrease in score representing improvement in stroke symptoms.
Symptomatic Intracerebral Hemorrhage (sICH) Rate | Within 7 days post-procedure
  Incidence of symptomatic intracerebral hemorrhage (sICH) in patients post-mechanical thrombectomy (MT), defined according to the European Cooperative Acute Stroke Study III (ECASS III) criteria. sICH is identified when there is:
  Imaging Evidence: Any intracerebral hemorrhage (ICH) detected on neuroimaging (computed tomography [CT] scan or magnetic resonance imaging [MRI]).
  Clinical Deterioration: A neurological worsening characterized by an increase of ≥4 points in the National Institutes of Health Stroke Scale (NIHSS) score from baseline or leading to death.
All-Cause Mortality at 90 Days | 90 days post-procedure
  Proportion of patients who have died from any cause by 90 days post-procedure.
Complication Rate | Immediately post-procedure up to 7 days
  Incidence of procedure-related complications (e.g., arterial dissection, vessel perforation).
Incremental Cost-Effectiveness Ratio (ICER) per Quality-Adjusted Life Year (QALY) Gained | From baseline (pre-procedure) through 90 days post-procedure, with economic modeling extended to a lifetime horizon (up to 20 years)
  The cost-effectiveness of mechanical thrombectomy (MT) compared to standard medical care (SMC) will be assessed by calculating the Incremental Cost-Effectiveness Ratio (ICER). This involves measuring both costs and health outcomes:
  Costs: Using hospital billing records and resource utilization data. Effectiveness: Measuring QALYs using the EQ-5D-5L questionnaire, a standardized instrument for measuring health outcomes.
  ICER Calculation: Explaining that the ICER will be calculated by dividing incremental costs by incremental QALYs.

CONTACTS AND LOCATIONS:
Overall Officials: ossama yassin MANSOUR, MD, PhD,, Principal Investigator — Alexandria University; farouk Hassan, MD,Phd, Principal Investigator — cairo university, Egypt; Atila Oscan Ozdimar, MD, PhD, Principal Investigator — Eskisehir Osmangazi University; Syed Irteza Hussain, MD, Principal Investigator — Cleveland Clinic Abu Dhabi; Faisal Alghamdi, MD, Principal Investigator — King Abdullah Medical City; Nadia Hammami, MD, Principal Investigator — institut National de Neurologie
Locations (1):
- Alexandria University Stroke network, Alexandria, Alexandria Governorate, Egypt